CLINICAL TRIAL: NCT00181792
Title: Family Risk Analysis of Substance Use in ADHD Youth Treated With Concerta
Brief Title: Family Risk Analysis of Substance Use in Attention Deficit Hyperactivity Disorder (ADHD) Youth Treated With Concerta
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paul Hammerness, MD, Assistant Professor Psychiatry, Massachusetts General Hospital
Other Study IDs: 2005-P-000278
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: ADHD; Smoking
Keywords: ADHD; smoking; familial risk
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Smoking

STUDY DESIGN:
Observational Model: Family Based
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The researchers will study 100 families over three years, each with a child (proband) between the ages of 12-17, with the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of ADHD. The researchers hypothesize smoking will be familial and ADHD probands with a family history of tobacco use will be at increased risk for early initiation and persistence of smoking, compared to ADHD probands with no family history of tobacco use.

DETAILED DESCRIPTION:
As Attention Deficit Hyperactivity Disorder (ADHD) is a documented risk factor for smoking in adolescents, and as theoretical considerations suggest that ADHD and tobacco use may share common underlying mechanisms, the proposed study looks to examine the association between smoking and ADHD. Since both ADHD and smoking are known to be familial disorders, one approach to examine the nature of the association between the two disorders is to conduct a familial risk analysis comparing ADHD youth who smoke and ADHD youth who don't smoke. Another approach is to conduct a genetic study, to identify candidate genes associated with nicotine abuse and dependence in ADHD youth and relatives.

This study includes:

1. assessment of psychopathology and substance use/dependence,
2. assessment of the family environment, and
3. assessment of molecular genetics in 100 families with at least one child (proband) between the ages of 12-17 with a DSM-IV diagnosis of ADHD.

ELIGIBILITY:
Inclusion Criteria:

* First-degree relative between the ages of 6-55 years of a family member (proband) between the ages of 12-17 with the DSM-IV diagnosis of ADHD

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: First-degree relative between the ages of 6-55 years of a family member (proband) between the ages of 12-17 with the DSM-IV diagnosis of ADHD
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2005-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hammerness, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States